CLINICAL TRIAL: NCT00120484
Title: Effect of Vitamin B12 on the Human Circadian Pacemaker
Brief Title: Effects of Vitamin B12 on the Body's Internal Clock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Jeanne F. Duffy, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT002571 (NIH); R21AT002571 (NIH)
Record Dates: First submitted 2005-07-13; First posted 2005-07-18 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Sleep Disorders, Circadian Rhythm
Keywords: Circadian Rhythm; Biological Clock; Complementary and Alternative Medicine
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vitamin B12

SUMMARY:
Circadian rhythms are 24-hour cycles that influence natural functions in the body such as heart rate, blood pressure, and body temperature. Circadian rhythms provide the body with an internal clock and affect sleep patterns. The purpose of this study is to determine the effects of vitamin B12 supplements on circadian rhythms and sleep-wake regulation.

DETAILED DESCRIPTION:
Individuals with circadian rhythm sleep disorder suffer from recurrent patterns of disrupted sleep that can significantly affect their daily functioning. Evidence suggests that vitamin B12 supplements may have a beneficial effect on sleep patterns. However, research on the effects of vitamin B12 supplements on sleep is limited. This study will determine the effects of vitamin B12 supplements on circadian rhythms and sleep-wake regulation.

This study will last 47 days. Participants will undergo a 3-week medical and psychological screening prior to study entry. Eligible participants will be admitted to the General Clinical Research Center where they will live in a private study room for the duration of the study. The room will be a time-free environment with no windows, clocks, television, or radio. Participants will not be able to make or receive telephone calls, and their bedtimes, wake times, and mealtimes will be determined by study researchers. Participants will be randomly assigned to receive three capsules of either vitamin B12 or placebo daily. Blood and saliva collection will occur daily to determine core body temperature and hormone levels. Performance tests to determine participants' cognitive abilities will be administered at regular intervals throughout each day. Participants' sleep will be recorded every night with polysomnography, which will monitor brain and muscle activity and breathing patterns during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of delayed sleep phase syndrome OR self-described as a "night owl"

Exclusion Criteria:

* History of medical illness
* History of psychiatric illness in participant or his or her family members
* Current medication or vitamin use
* Follow a vegan diet
* Significant visual problem
* Recent travel across time zones
* History of rotating shiftwork

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in circadian period | first 2 weeks vs. final 2 weeks of period assessments

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne F. Duffy, PhD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Harvard Medical School, Boston, Massachusetts, United States